CLINICAL TRIAL: NCT03446482
Title: Allocation of Physician Time in Anesthesiology Practice
Brief Title: Anesthesiology's Practice Time Evaluation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Principal Investigator, Vincent COMPERE, professor, University Hospital, Rouen
Other Study IDs: E2017-27
Record Dates: First submitted 2018-01-02; First posted 2018-02-26 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Anesthesiologist's Tasks

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observation of differents tasks — Evaluation by an external observer (nurse student in research stage or clinical research technician) of the distribution of medical time for the performance of the different tasks of anesthesiologist (in minutes)

SUMMARY:
The evolution of the health care system in Western countries has increased the scope of the tasks assigned to doctors in their daily lives. The burden of administrative tasks and the use of IT tools reduce the time spent with the patient. Indeed, in a very recent work published in the Annals of Internal Medicine, Sinsky et al. showed that in 4 different specialties (general medicine, internal medicine, cardiology and orthopaedics) for every hour spent in front of a patient, each physician spent two hours on tasks in the absence of the patient1. This distribution of time was found in the Wenger et al. study in 36 internal medicine interns, since a ratio of 1:3 between the working time spent in the presence of the patient (1.7 hours) and that spent in front of a computer (5.2 hours) was noted2.

The reduction in the clinical time devoted directly to the patient is a major source of dissatisfaction for physicians, which can even extend to burnout3. Moreover, it has been shown that the importance of computer tasks in everyday life is correlated with the occurrence of burnout4. Finally, beyond these clinical times directly or indirectly linked to patient care, the time spent on other tasks (administrative, travel time between different sites,...) appears to be significant (20% in Sinsky et al.)1.

The anesthesiologist faces the same constraints as other specialties, but no work has been specifically concerned with the distribution of time spent on the different tasks. Compared to other specialties, anesthesiologist is also regularly confronted with specific organisational tasks within the operating room that could reduce the time spent directly with patients.

The objective of this work is to determine the division of the different tasks in a anesthesiologist's work day by analysing the time spent directly with the patient but also that allocated to his or her care outside of his or her presence, as well as that devoted to organizational or administrative tasks.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiologist performing his day's work in an anaesthesia context
* Day including only clinical activity

Exclusion Criteria:

* Anesthesiologist isn't performing a day's work in an anaesthesia context
* Day not only includes clinical activity

Min Age: 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: anesthesiologist
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
time (minutes) of anesthesiologist's presence with the patient during anesthesia in operating room | 24 hours
  Evaluation by an external observer (nurse student in research internship or clinical research technician) of the time in minutes of anesthesiologist's presence with patient in operating room

SECONDARY OUTCOMES:
Satisfaction of the anesthesiologist on his workday Number/h of task's interruption | 3 days
  satisfaction was measured with numeric scale between 0 and 10

CONTACTS AND LOCATIONS:
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No